CLINICAL TRIAL: NCT07263672
Title: Clinical Efficacy of Local Anesthetic Agents With Interlaminar Epidural Steroid Injection for Chronic Neck Pain: A Prospective, Observational Study
Brief Title: Local Anesthetics in Cervical Epidural Injection
Status: Completed | Type: Observational
Sponsor: Mustafa Kurçaloğlu (Other)
Responsible Party: Sponsor-Investigator, Mustafa Kurçaloğlu, Assistant professor, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Other Study IDs: OMÜ KAEK 2021/300
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Chronic Neck Pain Due to Cervical Intervertebral Disc Herniation
Keywords: Pain; epidural; corticosteroid; local anesthetic; bupivacaine
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: Patients who received cervical epidural corticosteroid injection
- Group SLA: Patients who received cervical epidural corticosteroid and local anesthetic injection

SUMMARY:
This study aims to evaluate the efficacy of local anesthetic drugs in cervical epidural injections for chronic neck pain

DETAILED DESCRIPTION:
In this prospective observational study, patients were divided into two groups regarding the injected solution into the cervical epidural space. Group S received corticosteoroid injection and group LS received corticosteroid and bupivacaine injection. Pain severity scores (Numerical Rating Scale - NRS) and Neck Disability Index (NDI) scores were recored before the intervention and one, three, and six months after the interventions. Significant difference were searched between groups using by statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were planned to have a cervical epidural injection due to the pain originated from intervertebral disc herniation

Exclusion Criteria:

* Patients younger than18, those who were unwilling to participate, those who were pregnant or possibly pregnant, with infection or anatomic variations in the region of the procedure, allergic to the drugs to be used in the procedure and with coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic neck pain due to cervical intervertebral disc herniation and planned to have a cervical epidural injection due to the pain originated from intervertebral disc herniation
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | 6 months
  severity of pain from 0 to 11
Neck Disability Index (NDI) | 6 months
  an assessment tool for neck pain

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özkan, Professor, Principal Investigator — Ondokuz Mayis University Faculty of Medicine
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We agree to share participant data if there is a reasonable request from the reviewers or any kind of officials.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Aslan E, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagly N. The cultural adaptation, reliability and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2008 May 15;33(11):E362-5. doi: 10.1097/BRS.0b013e31817144e1. PMID 18469684

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT07263672/Prot_SAP_000.pdf
  • Informed Consent Form (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT07263672/ICF_001.pdf